CLINICAL TRIAL: NCT02668068
Title: A Multicenter, Randomized, Single-blind, Parallel-group Study of Combined Large Volume WLL With Clinical Grade Umbilical Cord Mesenchymal Stem Cells(MSC) Transplantation for Treatment of Pneumoconiosis
Brief Title: A Study on Pneumoconiosis Treated With Whole-lung Lavage Combined With Mesenchymal Stem Cells
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jianwu Dai (Other Government)
Collaborators: Southwest Hospital, China (Other); Nanjing Chest Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Jianwu Dai, Principal Investigator of Regenerative Medicine Laboratory, Institute of Genetics and Developmental Biology, CAS, Chinese Academy of Sciences
Organization: Chinese Academy of Sciences (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAS-XDA-SH/NCH/IGDB
Record Dates: First submitted 2016-01-20; First posted 2016-01-29 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2018-07

CONDITIONS: Pneumoconiosis
Keywords: Pneumoconiosis; Mesenchymal Stem Cells; whole-lung lavage (WLL)
MeSH Terms: conditions — Pneumoconiosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Active Comparator): Large volume whole-lung lavage (WLL) only
  Interventions: Procedure: large volume whole-lung lavage (WLL)
- Experimental Group (Experimental): Combined large volume WLL with clinical grade umbilical cord mesenchymal stem cells transplantation
  Interventions: Procedure: large volume whole-lung lavage (WLL); Biological: clinical grade umbilical cord mesenchymal stem cells

INTERVENTIONS:
Procedure: large volume whole-lung lavage (WLL) — Generally 1000 ~ 2000ml each time, 14 ~ 10 times totally, each side of the lung to 20 ~ 15 liters, until the lavage fluid from the black into a colorless clear clarification
Biological: clinical grade umbilical cord mesenchymal stem cells — 10^6 (1 million) /Kg/person cells of clinical grade umbilical cord MSCs will be injected after whole-lung lavage
  Arms: Experimental Group

SUMMARY:
Pneumoconiosis is a kind of lung disease due to inhalation of dust such as silica(common named Silicosis), coal and rock dust, characterized by inflammation, coughing, and fibrosis. Currently there is no effective drug treatment. The whole-lung lavage(WLL) can effectively clear the protein-like substances and inhaled dust deposited in the alveoli and bronchioles, as well as the pulmonary alveolar macrophage(PAM) and the resulting induced inflammation, fibrosis induced factor, serve to improve respiratory function, relieve symptoms of efficacy, but can't slow down or reverse the progression of pulmonary fibrosis.

By taking large volume whole-lung lavage (WLL) as a conventional therapy, this study intends to observe and evaluate the safety and efficiency of combined large volume WLL with mesenchymal stem cell (MSC) transplantation for treatment of Pneumoconiosis. Moreover, the immune regulation effect between large volume WLL and combined large volume WLL with MSC transplantation will also be preliminarily investigated and discussed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-70 years old.
2. Subjects had exposed to dusts with a long history.
3. Subjects with a clear clinical diagnosis to be silicotics or coal miners' pneumoconiosis patients.
4. Subjects with each detected index of pulmonary function test including FVC, FEV1 or MVV had exceeded 70% of the predicated value.
5. Subjects signed informed consent.

Exclusion Criteria:

1. Women of childbearing age at the stage of pregnancy or lactation, or those without taking effective contraceptive measures.
2. Subjects with syphilis or HIV positive antibody.
3. Subjects with infection aggravated within the past month.
4. Subjects suffering from any of the following pulmonary diseases: active tuberculosis, pulmonary embolism, pneumothorax, multiple huge bullae, uncontrolled asthma, severe pneumonia, acute exacerbation of chronic bronchitis, AECOPD, severe and / or extremely severe COPD, etc..
5. Subjects suffering from other serious diseases, such as myocardial infarction, unstable angina, cirrhosis, and acute glomerulonephritis.
6. Subjects suffering from other life-threatening diseases with an estimated life-span less than 2 years.
7. Subjects with leukopenia (WBC less than 4x109 / L) or agranulocytosis (WBC less than 1.5x109 / L or neutrophils less than 0.5x109 / L) caused by any reason.
8. Subjects with severe renal impairment, serum creatinine> 1.5 times the upper limit of normal.
9. Subjects with liver disease or liver damage: ALT, AST, total bilirubin> 2 times the upper limit of normal
10. Subjects with a history of mental illness or suicide risk, with a history of epilepsy or other central nervous system disorders.
11. Subjects with severe arrhythmias (such as ventricular tachycardia, frequent superventricular tachycardia, atrial fibrillation, and atrial flutter, etc.) or cardiac degree II or above conduction abnormalities displayed via 12-lead ECG.
12. Subjects with a history of alcohol or illicit drug abuse.
13. Subjects accepted by any other clinical trials within 3 months before the enrollment.
14. Subjects with poor compliance, difficult to complete the study.
15. Any other conditions that might increase the risk of subjects or interfere with the clinical trial.
16. Subjects accepted large volume whole-lung lavage treatment previously.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-01; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety Evaluation) | 6 months
  Clinical adverse events evaluated as definitely/ probably/possibly concerned with large volume lung lavage and / or mesenchymal stem cell therapy in this trial, and abnormal results of laboratory tests or other special examinations will be observed and recorded in detail.
Imaging indicator: Quantitative analysis of CT density histograms | 6 months after surgery

SECONDARY OUTCOMES:
Clinical Indicator 1: change in blood gas analysis | 6 months
  Including PH, PaCO2,PaO2, HCO3
Clinical Indicator 2: change in MRC chronic dyspnea scale | 6 months
Clinical Indicator 3: change in St. George's Respiratory Questionnaire (SGRQ) scale | 6 months
Immunological Indicator in serum : response level of CD4+ T lymphocyte subsets (Th1/Th2/Th17) | 6 months
Immunological Indicator in lavage fluid : response level of CD4+ T lymphocyte subsets (Th1/Th2/Th17) | 6 months
Immunological Indicator in serum : expression levels of various cytokines including TNF-α, IL1-β, MIP-1α, TIMP1, PDGF | 6 months
Immunological Indicator in lavage fluid: expression levels of various cytokines including TNF-α, IL1-β, MIP-1α, TIMP1, PDGF | 6 months
Fibrosis Indicators in serum: expression levels of TGF-β1, hydroxyproline, MMP2, MMP9 | 6 months
Fibrosis Indicators in lavage fluid: expression levels of TGF-β1, hydroxyproline, MMP2, MMP9 | 6 months
self-evaluation | 6 months
  Self-evaluation will be also classified into four levels: effective, improved, stable and invalid

CONTACTS AND LOCATIONS:
Overall Officials: JianWu Dai, Ph.D, Principal Investigator — Chinese Academy of Sciences; Wei Xiong, M.D, Study Chair — First Affiliated Hospital of the Third Military University, PLA (Southwest Hospital); Xiaotian Dai,, M.M, Study Director — First Affiliated Hospital of the Third Military University, PLA (Southwest Hospital); Yingming Zhang, M.M, Study Director — Nanjing Chest Hospital; Shencun Fang, M.M, Study Director — Nanjing Chest Hospital
Locations (2):
- China (2):
  - First Affiliated Hospital of the Third Military University, PLA (Southwest Hospital), Chongqing, Chongqing Municipality
  - Nanjing Chest Hosptial, Nanjing, Jiangsu